CLINICAL TRIAL: NCT02736058
Title: Surgical Classification of Abnormal Placentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Hussein, Lecturer of Obstetrics and Gynecology, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PP2202016
Record Dates: First submitted 2016-02-22; First posted 2016-04-13 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Adherent Placenta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Participants (Experimental): the included pregnant females will undergo trans-abdominal sonography as well as trans-vaginal sonography , to diagnose the abnormal placentation and the results will be compared to the intra- operative as well as the pathological examination of the specimen.
  Interventions: Device: Trans- abdominal sonography; Device: Trans-vaginal sonography; Procedure: post-operative pathological specimen examination

INTERVENTIONS:
Device: Trans- abdominal sonography
Device: Trans-vaginal sonography
Procedure: post-operative pathological specimen examination

SUMMARY:
Reaching the proper pre-operative diagnosis for abnormal placentation in crucial to markedly decrease the intra-operative complications as well as the maternal morbidity and mortality. In this trial researchers aim to set up some pre-operative sonographic criteria that would help in planning the surgical procedure as well as setting up a surgical classification for the abnormally adherent placenta.

ELIGIBILITY:
Inclusion Criteria:

* abnormal placental site (placenta previa)

Exclusion Criteria:

* refusal to participate in the study
* cases with normal placental location ( fundal, anterior or posterior wall not reaching the lower uterine segment)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Hussein, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided